CLINICAL TRIAL: NCT06223009
Title: A First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Examine the Safety, Tolerability, and Pharmacokinetics of cNP8 in Healthy Adults
Brief Title: Phase 1 Healthy Volunteer Burn Therapy Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neomatrix Therapeutics, Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NMT-cNP8-101; HT9425-23-1-1064 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single ascending doses of cNP8 (Experimental): Subjects will be randomized to receive either a single dose of cNP8 or placebo (6:2). The doses will be studied sequentially starting with the lowest cNP8 dose.
  Interventions: Drug: cNP8
- Single doses of placebo administered (Placebo Comparator): Subjects will be randomized to receive either a single dose of cNP8 or placebo (6:2).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: cNP8 — cNP8 for injection is provided as a sterile lyophilizate for solution for infusion. Subjects will receive a single 30 minute IV infusion of cNP8 at their assigned dose.
  Arms: Single ascending doses of cNP8
Other: Placebo — Subjects not randomized to cNP8 will receive a single 30 minute IV infusion of placebo.
  Arms: Single doses of placebo administered

SUMMARY:
This is a Phase 1, single-center, randomized, double-blind, placebo-controlled, first-in-human study to evaluate the safety of an investigational drug to treat burns. Participants will be healthy male and female adults. The study will consist of a screening period, inpatient dosing and observation period and safety follow-up. Participants will receive 1 intravenous dose of the investigational drug or placebo. Duration of participation will be approximately 38 days, which includes a maximum of a 30 day screening period and a study period of approximately 8 days.

DETAILED DESCRIPTION:
Up to 32 healthy, male and female subjects will be enrolled in this Phase 1, single-center, randomized, double-blind, placebo-controlled, first-in-human study. Eligible subjects will be confined to a Phase 1 unit for approximately 48 hours and receive a one time IV dose of study medication. They will be required to return for a safety follow-up visit one week later.

Doses will be studied sequentially starting with the lowest dose of the investigational drug, cNP8. Each dose cohort will include a total of 6 subjects dosed with cNP8 and 2 subjects dosed with placebo.

A sentinel dosing plan with staggered enrollment will be employed. For each dosing cohort, 2 subjects will be dosed (1 with cNP8 and 1 with placebo) and monitored for serious and/or severe adverse events (AEs). If no serious or severe AEs occur in 24 hours postdose, the remaining 6 subjects in the cohort will be dosed.

Safety evaluations, including laboratory tests, vital sign measurements and electrocardiograms, will be performed at several timepoints throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 kg/m2 to 32 kg/m2 and body weight of greater than or equal to 50 kg.
* Use of highly-effective methods of birth control
* Willing and able to remain in a clinical research unit for the required study duration and return for the outpatient visit

Exclusion Criteria:

* A clinically significant laboratory abnormality or other finding indicative of a clinically-significant exclusionary disease
* A history of asymptomatic or mild COVID within 30 days of study drug administration
* A history of hospitalization with COVID within 6 months prior to study drug administration
* A history of COVID vaccination within 1 month prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events from dosing through follow-up | Day -1, Day 2, Day 8 Safety Follow-up
  Clinical safety laboratory data will be collected
Incidence and severity of adverse events from dosing through follow-up | Day -1, 1 hour postdose, 6 hours postdose, Day 2 and Day 8 Safety Follow-up
  Electrocardiograms will be performed
Incidence and severity of adverse events from dosing through follow-up | Predose, 0.25,0.50, 0.75,1,1.5, 2,4,6,12 hours postdose, Day 2 and Day 8 Safety Follow-up
  Vital signs

SECONDARY OUTCOMES:
Pharmacokinetic profile | Predose, 0.25,0.50,0.75,1,1.5, 2,4,6,12 hours postdose
  Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Saint Paul, Minnesota, United States